CLINICAL TRIAL: NCT02414815
Title: Reverse Prediction of Ion Channel Remodeling in Patients With Atrial Fibrillation Utilizing Monophasic Action Potential and Mathematical Modeling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 4-2014-0685
Record Dates: First submitted 2015-04-03; First posted 2015-04-13 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheters

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AF group (Experimental): Atrial fibrillation
  Interventions: Device: Monophasic action potential(MAP) catheter

INTERVENTIONS:
Device: Monophasic action potential(MAP) catheter — After ordinary procedure for electrophysiologic study or catheter ablation, the investigators will replace conventional catheter to monophasic action potential (MAP) recording catheter through right femoral sheath. MAP recording catheter is introduced to endocardial surface of atrium, and we record atrial MAP at variable pacing cycle lengths: steady state cycle lengths of 600, 400, 300, 240, 220, 240, 260, 300, 400 and 600 ms. At each cycle length, pacing was applied for 20 sec. It takes less than 5 min to acquire MAP recordings.

SUMMARY:
Atrial fibrillation(AF) is the most common sustained arrhythmia in humans. The loss of rate-dependent action potential duration(APD) adaptation is one of the characteristics of atrial fibrillation, but detailed understanding of mechanism is limited. Thus, we propose to utilize the monophasic action potential recording data from human patients in three groups, control, paroxysmal and persistent atrial fibrillation, and apply reverse engineering method to quantify the extent of electrical remodeling of ionic channel parameters using a mathematical model of atrial cell. Our approach will be useful in developing drug targets for ion channels in atrial fibrillation patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients agreement of consent
* AF patient age 19-75
* Patients who undergoing catheter ablation of atrial fibrillation or supraventricular tachycardia
* Patient agreement of consent who admission for catheter ablation

Exclusion Criteria:

* Patients who do not agree with study inclusion
* Permanent AF refractory to electrical cardioversion
* AF with rheumatic valvular disease
* Patients with left atrial diameter greater than 60mm
* Patients with age less than 19 or more 75

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-08-28; Primary Completion 2017-03-02 (Actual); Study Completion 2017-03-02 (Actual)

PRIMARY OUTCOMES:
Recurrence of AF | One year after the last enrollment
  The investigators will acquire monophasic action potential from patient's atrium. Then, we will estimate cardiac ion current status of the patients by reverse engineering and computer simulation. The patients will be followed up longer than 12 months based on 2012 ACC/AHA/ESC guidelines. Primary outcomes of the study are AF recurrence and antiarrhythmic drug sensitivity. Those data will be counted and compared with the patient's own ion current status deducted by simulation study with monophasic action potentials.
Antiarrhythmic drug sensitivity | One year after the last enrollment
  The investigators will acquire monophasic action potential from patient's atrium. Then, we will estimate cardiac ion current status of the patients by reverse engineering and computer simulation. The patients will be followed up longer than 12 months based on 2012 ACC/AHA/ESC guidelines. Primary outcomes of the study are AF recurrence and antiarrhythmic drug sensitivity. Those data will be counted and compared with the patient's own ion current status deducted by simulation study with monophasic action potentials.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Cardiovascular Hospital, Yonsei University Health System, Seoul, South Korea